CLINICAL TRIAL: NCT00952653
Title: An Open-Label, Two-Period, Sequential Drug Interaction Study to Evaluate the Effect of Multiple Doses of Desvenlafaxine Succinate Sustained Release (DVS SR) on the Pharmacokinetics of Midazolam When Coadministered in Healthy Subjects
Brief Title: Study Evaluating the Effect of Desvenlafaxine on the Pharmacokinetics of Midazolam
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3151A1-1205; B2061001
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Results first posted 2011-08-02 (Estimated); Last update posted 2011-08-15 (Estimated); Status verified 2011-08

CONDITIONS: Major Depressive Disorder
Keywords: depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DVS SR (Experimental)
  Interventions: Drug: Desvenlafaxine Succinate Sustained Release; Drug: Midazolam

INTERVENTIONS:
Drug: Desvenlafaxine Succinate Sustained Release — 50 mg DVS SR tablet days 1-6, period 2 only.
Drug: Midazolam — 4 mg midazolam (2 mL midazolam syrup) day 1, period 1 and day 6, period 2.

SUMMARY:
The main purpose of this study is to evaluate the effect of desvenlafaxine administered as DVS SR on the pharmacokinetics of midazolam in healthy male and female subjects. The amount of drug in the body and the effect of the drug will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Men or non-pregnant, non-lactating women, 18 to 55 years of age inclusive at screening.
* Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12-lead electrocardiogram (ECG).
* Nonsmoker or smoker of fewer than 10 cigarettes per day as determined by history.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 Ilbs).

Exclusion Criteria:

* Presence or history of any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
* Presence or history of glaucoma or intraocular pressure.
* Any surgical or medical condition that may interfere with the absorption, distribution, metabolism, or excretion of the investigational product.
* Allergy to midazolam, other benzodiazepine, desvenlafaxine, or venlafaxine.
* Acute disease state (eg, nausea, vomiting, fever, or diarrhea) with 7 days before study day 1.
* Admitted alcohol abuse or history of alcohol use that may interfere with the subject's ability to comply with the protocol requirements. History of drug abuse within 1 year before study day 1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2010-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3151A1-1205&StudyName=Study%20Evaluating%20the%20Effect%20of%20Desvenlafaxine%20on%20the%20Pharmacokinetics%20of%20Midazolam

RESULTS

PARTICIPANT FLOW:
Groups:
- DVS SR 50 mg, Midazolam 4 mg: Midazolam (MDZ) 4 milligram (mg) syrup (2 mg per milliliter [mg/mL]) as a single oral dose Period 1 / Day 1. Desvenlafaxine sustained-release formulation (DVS SR) 50 mg tablet as a single oral dose Period 2 / Day 1 to Day 5 (steady state); DVS SR 50 mg tablet as a single oral dose and midazolam 4 mg syrup (2 mg/mL) as a single oral dose Period 2 / Day 6.
Period: Period 1: MDZ Alone
Arm/Group | DVS SR 50 mg, Midazolam 4 mg
Started | 28
Completed | 28
Not Completed | 0
Period: Period 2: Coadministration DVS SR, MDZ
Arm/Group | DVS SR 50 mg, Midazolam 4 mg
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- DVS SR 50 mg, Midazolam 4 mg: Midazolam 4 mg syrup (2 mg/mL) as a single oral dose Period 1 / Day 1. DVS SR 50 mg tablet as a single oral dose Period 2 / Day 1 to Day 5 (steady state); DVS SR 50 mg tablet as a single oral dose and midazolam 4 mg syrup (2 mg/mL) as a single oral dose Period 2 / Day 6.
Arm/Group | DVS SR 50 mg, Midazolam 4 mg
Number analyzed (Participants) | 28
Age, Customized [Number; unit: participants]
  18 to 25 years | 2
  26 to 35 years | 9
  36 to 45 years | 13
  > 45 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Midazolam Area Under the Plasma Concentration-time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) Following Midazolam Alone and When Coadministered With DVS SR
Description: AUCinf measured as nanograms multiplied by hours divided by milliliters (ng*hr/mL).
Time Frame: Period 1 / Day 1 and Period 2 / Day 6: 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, and 24 hours following dosing
Population: PK parameter analysis population: all enrolled and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period. N=number of participants contributing to the mean.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Midazolam 4 mg (Period 1): Midazolam 4 mg syrup (2 mg/mL) as a single oral dose Period 1 / Day 1.
- DVS SR 50 mg, Midazolam 4 mg (Period 2): DVS SR 50 mg tablet as a single oral dose Period 2 / Day 1 to Day 5 (steady state); DVS SR 50 mg tablet as a single oral dose and midazolam 4 mg syrup (2 mg/mL) as a single oral dose Period 2 / Day 6.
Arm/Group | Midazolam 4 mg (Period 1) | DVS SR 50 mg, Midazolam 4 mg (Period 2)
Number analyzed (Participants) | 26 | 25
ng*hr/mL | 54.69 (26.670) | 39.45 (13.301)
Statistical Analysis 1: Comparison: Midazolam 4 mg (Period 1) vs DVS SR 50 mg, Midazolam 4 mg (Period 2); DVS SR + Midazolam (test) versus Midazolam (reference). Based on the sample size, this study has at least 85% power overall to demonstrate the lack of an interaction [that is, equivalence in both AUCinf and Cmax and both midazolam and 1-hydroxy midazolam], where overall study power is to be based on the product of the individual powers of the parameters of interest; Test type: Superiority or Other; ratio of adjusted geometric means = 71.40, 90% CI 2-sided [65.08 to 78.33] — Values have been back-transformed from the log scale

2. Primary Outcome: Midazolam Maximum Observed Plasma Concentration (Cmax) Following Midazolam Alone and When Coadministered With DVS SR
Description: Cmax measured as nanograms per milliliters (ng/mL).
Time Frame: as for outcome 1
Population: PK parameter analysis population; N=number of participants contributing to the mean.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Midazolam 4 mg (Period 1) | DVS SR 50 mg, Midazolam 4 mg (Period 2)
Number analyzed (Participants) | 26 | 26
ng/mL | 21.20 (7.1216) | 18.24 (5.1116)
Statistical Analysis 1: Comparison: Midazolam 4 mg (Period 1) vs DVS SR 50 mg, Midazolam 4 mg (Period 2); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio of adjusted geometric means = 86.08, 90% CI 2-sided [79.04 to 93.74] — Values have been back-transformed from the log scale

3. Primary Outcome: 1-Hydroxy-Midazolam (Analyte) Area Under the Plasma Concentration-time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) Following Midazolam Alone and When Coadministered With DVS SR
Description: 1-Hydroxy-Midazolam is an analyte of Midazolam.
Time Frame: as for outcome 1
Population: PK parameter analysis population; N=number of participants contributing to the mean.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Midazolam 4 mg (Period 1) | DVS SR 50 mg, Midazolam 4 mg (Period 2)
Number analyzed (Participants) | 26 | 26
ng*hr/mL | 36.87 (28.230) | 30.74 (14.649)
Statistical Analysis 1: Comparison: Midazolam 4 mg (Period 1) vs DVS SR 50 mg, Midazolam 4 mg (Period 2); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio of adjusted geometric means = 92.55, 90% CI 2-sided [87.43 to 97.97] — Values have been back-transformed from the log scale

4. Primary Outcome: 1-Hydroxy-Midazolam (Analyte) Maximum Observed Plasma Concentration (Cmax) Following Midazolam Alone and When Coadministered With DVS SR
Time Frame: as for outcome 1
Population: PK parameter analysis population; N=number of participants contributing to the mean.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Midazolam 4 mg (Period 1) | DVS SR 50 mg, Midazolam 4 mg (Period 2)
Number analyzed (Participants) | 26 | 26
ng/mL | 14.93 (6.5282) | 15.10 (6.2472)
Statistical Analysis 1: Comparison: Midazolam 4 mg (Period 1) vs DVS SR 50 mg, Midazolam 4 mg (Period 2); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio of adjusted geometric means = 101.17, 90% CI 2-sided [92.96 to 110.11] — Values have been back-transformed from the log scale

5. Secondary Outcome: Midazolam Area Under the Plasma Concentration-time Profile From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) Following Midazolam Alone and When Coadministered With DVS SR
Time Frame: as for outcome 1
Population: PK parameter analysis population; N=number of participants contributing to the mean.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Midazolam 4 mg (Period 1) | DVS SR 50 mg, Midazolam 4 mg (Period 2)
Number analyzed (Participants) | 26 | 26
ng*hr/mL | 52.85 (23.980) | 38.11 (12.522)
Statistical Analysis 1: Comparison: Midazolam 4 mg (Period 1) vs DVS SR 50 mg, Midazolam 4 mg (Period 2); DVS SR + Midazolam (test) versus Midazolam (reference); Test type: Superiority or Other; ratio of adjusted geometric means = 72.10, 90% CI 2-sided [66.04 to 78.72] — Values have been back-transformed from the log scale

6. Secondary Outcome: Midazolam Time to Cmax (Tmax) Following Midazolam Alone and When Coadministered With DVS SR
Time Frame: as for outcome 1
Population: PK parameter analysis population; N=number of participants contributing to the median.
Measure: Median (Full Range); unit: hr
Arm/Group | Midazolam 4 mg (Period 1) | DVS SR 50 mg, Midazolam 4 mg (Period 2)
Number analyzed (Participants) | 26 | 26
hr | 0.517 [0.250 to 1.50] | 0.500 [0.250 to 1.02]

7. Secondary Outcome: Midazolam Terminal Half-life (t 1/2) Following Midazolam Alone and When Coadministered With DVS SR
Time Frame: as for outcome 1
Population: PK parameter analysis population; N=number of participants contributing to the mean.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Midazolam 4 mg (Period 1) | DVS SR 50 mg, Midazolam 4 mg (Period 2)
Number analyzed (Participants) | 26 | 25
hr | 5.320 (1.5948) | 4.648 (1.7436)

8. Secondary Outcome: 1-Hydroxy-Midazolam (Analyte) Area Under the Plasma Concentration-time Profile From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) Following Midazolam Alone and When Coadministered With DVS SR
Time Frame: as for outcome 1
Population: PK parameter analysis population; N=number of participants contributing to the mean.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Midazolam 4 mg (Period 1) | DVS SR 50 mg, Midazolam 4 mg (Period 2)
Number analyzed (Participants) | 26 | 26
ng*hr/mL | 37.09 (25.371) | 32.42 (14.881)
Statistical Analysis 1: Comparison: Midazolam 4 mg (Period 1) vs DVS SR 50 mg, Midazolam 4 mg (Period 2); DVS SR + Midazolam (test) versus Midazolam (reference); Test type: Superiority or Other; ratio of adjusted geometric means = 87.39, 90% CI 2-sided [80.42 to 94.96] — Values have been back-transformed from the log scale

9. Secondary Outcome: 1-Hydroxy-Midazolam (Analyte) Time to Cmax (Tmax) Following Midazolam Alone and When Coadministered With DVS SR
Time Frame: as for outcome 1
Population: PK parameter analysis population; N=number of participants contributing to the median.
Measure: Median (Full Range); unit: hr
Arm/Group | Midazolam 4 mg (Period 1) | DVS SR 50 mg, Midazolam 4 mg (Period 2)
Number analyzed (Participants) | 26 | 26
hr | 1.00 [0.250 to 1.50] | 0.500 [0.250 to 1.02]

10. Secondary Outcome: 1-Hydroxy-Midazolam (Analyte) Terminal Half-life (t 1/2) Following Midazolam Alone and When Coadministered With DVS SR
Time Frame: as for outcome 1
Population: PK parameter analysis population; N=number of participants contributing to the mean.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Midazolam 4 mg (Period 1) | DVS SR 50 mg, Midazolam 4 mg (Period 2)
Number analyzed (Participants) | 21 | 20
hr | 5.396 (2.0638) | 4.616 (1.7976)

ADVERSE EVENTS:
Time Frame: Baseline up to Period 2 / Day 7 final visit (Adverse Events) or up to 28 days after last study treatment (Serious Adverse Events)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study. Participants are counted for each treatment sequence.
Groups:
- DVS SR 50 mg (Period 2 / Day 1 to Day 5): DVS SR 50 mg tablet as a single oral dose Period 2 / Day 1 to Day 5 (steady state).
- DVS SR 50 mg + Midazolam 4 mg (Period 2 / Day 6): DVS SR 50 mg tablet as a single oral dose and midazolam 4 mg syrup (2 mg/mL) as a single oral dose Period 2 / Day 6.
Arm/Group | Midazolam 4 mg (Period 1) | DVS SR 50 mg (Period 2 / Day 1 to Day 5) | DVS SR 50 mg + Midazolam 4 mg (Period 2 / Day 6)
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 21/28 | 16/28 | 24/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Midazolam 4 mg (Period 1) (N=28) | DVS SR 50 mg (Period 2 / Day 1 to Day 5) (N=28) | DVS SR 50 mg + Midazolam 4 mg (Period 2 / Day 6) (N=28)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 4 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 3 | 4
Feeling abnormal (General disorders) | 0 | 2 | 0
Feeling of relaxation (General disorders) | 1 | 0 | 0
Hunger (General disorders) | 0 | 1 | 1
Thirst (General disorders) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 6 | 1
Hypersomnia (Nervous system disorders) | 0 | 1 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 20 | 0 | 20
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 3 | 1
Middle insomnia (Psychiatric disorders) | 0 | 1 | 0
Urine flow decreased (Renal and urinary disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.